CLINICAL TRIAL: NCT01539863
Title: Chiropractic Maintenance Care of Persistent or Recurrent Low Back Pain. A Randomized Controlled Trial With 1 Year Follow up
Brief Title: Chiropractic Maintenance Care of Persistent or Recurrent Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Iben Axen, Principal Investigator, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: KIIMMIIR
Record Dates: First submitted 2012-02-22; First posted 2012-02-28 (Estimated); Results first posted 2021-03-12 (Actual); Last update posted 2023-10-16 (Actual); Status verified 2023-10

CONDITIONS: Recurrent Low Back Pain; Persistent Low Back Pain; Chronic Low Back Pain
MeSH Terms: conditions — Low Back Pain | interventions — Long-Term Care; Therapeutics; Health Services Needs and Demand

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment at regular intervals (Experimental): Participants will be scheduled to receive the intervention, maintenance care, i.e. care on a regular basis throughout the study period.Care may consist of manual treatment but also of e.g. advice concerning exercises, ergonomic adaptation and stress management
  Interventions: Other: maintenance care
- Treatment as needed (Active Comparator): Participants will receivethe intervention, i.e.care only when requested by them, i.e. when experiencing a relapse or deterioration
  Interventions: Other: Treatment as needed

INTERVENTIONS:
Other: maintenance care — Participants will receive treatment at regular intervals during the study, a maximum of 12 and a minimum of 4 treatments as decided by the treating chiropractor
  Arms: Treatment at regular intervals
Other: Treatment as needed — Participants may never receive treatment, there is no upper limit
  Arms: Treatment as needed

SUMMARY:
As low back pain is often a recurrent and sometime persistent problem, research into prevention is important. Chiropractors have traditionally treated patients with maintenance care, which means that patients are seen on a regular basis to prevent recurrences or to stop a persistent problem getting worse. However, it is not known if this has the expected effect.

This study will test the effectiveness of the maintenance care approach. Patients with recurrent or persistent low back pain will be treated in accordance with two different models. The first model is the maintenance care model, meaning that chiropractors will see the patient on a regular basis, regardless symptoms. The other model means that patients should be treated patients only when they themselves experience symptoms bad enough to seek care. After one year, it will be possible to see if there has been any difference between the groups in terms of pain, disability, quality of life and total number of treatments over the study period and to investigate if there is any difference in the cost-effectiveness between the two treatment models.Thus, the study hypothesis is that there is no difference between the two models regarding the number of days with pain.

This study will be a multi-centre trial, and as part of the study, it will be necessary to formalize a network of research clinics all over Sweden in which participating chiropractors accept to perform complex data collection. This network will then have the expertise and potential to perform future clinical studies together with networks in other countries, allowing large clinical trials across countries.

ELIGIBILITY:
Inclusion Criteria:

* non-specific low back pain > 30 days previous year
* non-specific low back pain with previous episodes
* age 18-65
* access to a mobile phone
* knowledge of how to text message
* proficiency in the Swedish language
* must rate themselves as "definitely improved" by the 4th visit

Exclusion Criteria:

* pregnancy
* contraindication to spinal manipulative therapy
* liability issues

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 328 (Actual)
Dates: Start 2012-03; Primary Completion 2016-08 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Irene Jensen, PhD, Study Director — Karolinska Institutet
Locations (1):
- Karolinska Institutet, Stockholm, Sweden

REFERENCES:
- [Derived] Eklund A, Palmgren PJ, Jakobsson U, Axen I. Development and evaluation of the MAINTAIN instrument, selecting patients suitable for secondary or tertiary preventive manual care: the Nordic maintenance care program. Chiropr Man Therap. 2022 Mar 17;30(1):15. doi: 10.1186/s12998-022-00424-6. PMID 35300729
- [Derived] Eklund A, Hagberg J, Jensen I, Leboeuf-Yde C, Kongsted A, Lovgren P, Jonsson M, Petersen-Klingberg J, Calvert C, Axen I. The Nordic maintenance care program: maintenance care reduces the number of days with pain in acute episodes and increases the length of pain free periods for dysfunctional patients with recurrent and persistent low back pain - a secondary analysis of a pragmatic randomized controlled trial. Chiropr Man Therap. 2020 Apr 21;28(1):19. doi: 10.1186/s12998-020-00309-6. PMID 32316995
- [Derived] Eklund A, Bergstrom G, Bodin L, Axen I. Do psychological and behavioral factors classified by the West Haven-Yale Multidimensional Pain Inventory (Swedish version) predict the early clinical course of low back pain in patients receiving chiropractic care? BMC Musculoskelet Disord. 2016 Feb 12;17:75. doi: 10.1186/s12891-016-0933-y. PMID 26867930
- [Derived] Eklund A, Bergstrom G, Bodin L, Axen I. Psychological and behavioral differences between low back pain populations: a comparative analysis of chiropractic, primary and secondary care patients. BMC Musculoskelet Disord. 2015 Oct 19;16:306. doi: 10.1186/s12891-015-0753-5. PMID 26483193
- [Derived] Eklund A, Axen I, Kongsted A, Lohela-Karlsson M, Leboeuf-Yde C, Jensen I. Prevention of low back pain: effect, cost-effectiveness, and cost-utility of maintenance care - study protocol for a randomized clinical trial. Trials. 2014 Apr 2;15:102. doi: 10.1186/1745-6215-15-102. PMID 24690201

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with persistent or recurrent LBP were screened for eligibility in a stepwise manner (at Baseline 1, Baseline 2 and inclusion visit). The study started at the inclusion visit, when the initial treatment plan was completed when the clinician perceived that the patient's next visit could be scheduled with an interval of 1 month or longer, at which patients were randomly allocated to one of the treatment arms. Recruitment lasted from 2012 to 2016, in 40 Swedish chiropractic clinics.
Pre-assignment Details: Some individuals were lost in the inclusion process: At the 4th visit (baseline 2) a total of 616 subjects were screened for definite improvement, where 176 subjects were excluded from the trial. At the inclusion visit, 328 subjects were randomized into the trial, thus another 112 subjects were lost for unknown reasons.
Period: Overall Study
Arm/Group | Treatment at Regular Intervals | Treatment as Needed
Started | 166 | 162
Completed | 161 | 158
Not Completed | 5 | 4
Not completed — Lost to Follow-up | 5 | 4

BASELINE CHARACTERISTICS:
Population: Four individuals declined participation after randomization
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment at Regular Intervals | Treatment as Needed | Total
Number analyzed (Participants) | 164 | 160 | 324
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: 4 individuals declined participation after randomization
  years | 43.4 (11.7) | 43.0 (13.1) | 43.3 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Information about gender was not available for all subjects
  Participants
    number analyzed (Participants) | 150 | 141 | 291
    Female | 96 | 85 | 181
    Male | 54 | 56 | 110
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Sweden | 164 | 160 | 324

OUTCOME MEASURES:

1. Primary Outcome: Number of Days With Bothersome Low Back Pain
Description: Participants will report their number of days with bothersome low back pain via text message (SMS) on a weekly basis for 52 weeks.
Time Frame: 12 months
Measure: Mean (95% Confidence Interval); unit: Number of days with bothersome pain
Arm/Group | Treatment at Regular Intervals | Treatment as Needed
Number analyzed (Participants) | 161 | 158
Number of days with bothersome pain | 85.2 [83.5 to 87.0] | 98 [95.9 to 100.1]

2. Secondary Outcome: Cost-effectiveness
Description: Cost-effectiveness will be based on Quality Adjusted Life Years calculated through the use of the Euroqol-5 instrument, these results are not yet published
Time Frame: 12 months
Reporting Status: Not Posted, anticipated posting 2024-11

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Treatment at Regular Intervals | Treatment as Needed
All-Cause Mortality (participants affected / at risk) | 0/164 | 0/160
Serious Adverse Events (participants affected / at risk) | 0/164 | 0/160
Other Adverse Events (participants affected / at risk) | 43/164 | 40/160
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment at Regular Intervals (N=164) | Treatment as Needed (N=160)
Minor (Musculoskeletal and connective tissue disorders) | 43 (43) | 40 (40) — Local soreness Felt tired

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No